CLINICAL TRIAL: NCT06950034
Title: A Phase 1, Open-Label, Dose Escalation and Expansion Study of STX-0712 in Patients With Advanced Hematologic Malignancies
Brief Title: A Phase 1 Study of STX-0712 in Patients With Advanced Hematological Malignancies (CMML and AML)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Solu Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SOLU-ONC-001
Record Dates: First submitted 2025-04-09; First posted 2025-04-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Myelomonocytic Leukemia; Chronic Myelomonocytic Leukemia (CMML); Chronic Myelomonocytic Leukemia-1; Chronic Myelomonocytic Leukemia-2; Refractory Chronic Myelomonocytic Leukemia; CMML; Acute Myeloid Leukemia; Acute Myeloid Leukemia (AML); Acute Myeloid Leukemia Post Cytotoxic Therapy; Acute Myeloid Leukemias; Refractory Acute Myeloid Leukemia (AML); Acute Monocytic Leukemia
Keywords: refractory/resistant CMML; CMML; AML; monocytic AML; Relapsed/refractory AML; monocytic-predominant AML; Chronic Myelomonocytic Leukemia; Acute Myeloid Leukemia; Refractory Chronic Myelomonocytic Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute; Leukemia, Monocytic, Acute

STUDY DESIGN:
Intervention Model Description: This is a Dose Escalation and Dose expansion study testing STX-0712 in 2 indications: CMML (Cohort 1) and Monocytic and/or monocytic predominant AML (Cohort 2).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation in CMML Patients (Experimental): STX-0712 will be administered every 21 days.
  Interventions: Biological: STX-0712
- Dose Escalation in AML Patients (Experimental): STX-0712 will be administered every 21 days.
  Interventions: Biological: STX-0712
- Dose Expansion in CMML (Experimental): STX-0712 will be administered every 21 days.
  Interventions: Biological: STX-0712
- Dose Expansion in AML (Experimental): STX-0712 will be administered every 21 days.
  Interventions: Biological: STX-0712

INTERVENTIONS:
Biological: STX-0712 — STX-0712 is IV administered every 21 days until the patient discontinues treatment.

SUMMARY:
This is a first-in-human, multicenter, open-label, phase 1 study to evaluate the safety, PK, PD and preliminary efficacy of STX-0712 in patients with advanced CMML and AML for whom there are no further treatment options known to confer clinical benefit.

DETAILED DESCRIPTION:
This is an open-label, non-randomized phase 1 trial to assess the safety and preliminary efficacy of STX-0712 in refractory/resistant CMML and relapsed/refractory monocytic or monocytic-predominant AML. The study will be conducted in two parts: Dose Escalation (Part 1) and Dose Expansion (Part 2). Dose Escalation will accrue CMML and AML patients across 2 cohorts using the BOIN adaptive design, followed by Dose Expansion in both cohorts using Simon's 2-Stage Design. Cohort 1 will enroll approximately 3-6 CMML patients at each dose level. After at least two dose levels have been deemed safe in Cohort 1, the Sponsor may decide to open Cohort 2 to enroll AML patients. Approximately 20 patients will be enrolled in each Dose Expansion cohort. All eligible participants will be administered the study drug, STX-0712, as a single intravenous (IV) infusion every 21 days. Patients will remain on study therapy until treatment discontinuation criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Refractory/resistant CMML, defined as: Diagnosis of CMML 1 or 2; and has not responded to at least 4 cycles of hypomethylating agents (HMAs)(for myeloproliferative CMML - HMAs or hydroxyurea) or discontinued prior to 4 cycles due to toxicity or has progressive disease OR
* Relapsed/refractory monocytic or monocytic predominant AML. Monocytic predominant AML is defined as ≥50% monocytes and/or monocytic precursors (promonocytes/monoblasts) and expressing at least two monocytic markers including CD4, CD11c, CD14, CD36, or CD64; and peripheral blood white blood cell (WBC) <30,000/µL (microliters) and <20% circulating blasts.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2.
* Life expectancy of >2 months and stable enough to complete two cycles of STX-0712, in the opinion of the Investigator.
* Adequate organ function.
* Both females of child-bearing potential and males must agree to use acceptable contraceptive methods for the duration of time in the study and to continue to use acceptable contraceptive methods for 90 days after last STX-0712 infusion.
* Able to understand and willing to sign a written informed consent form.
* Willing and able to comply with study procedures and follow-up examinations.

Exclusion Criteria:

* Has any of the following disease-specific conditions: For CMML: Myelodysplastic syndrome/myeloproliferative neoplasm (MDS/MPN) overlap syndromes other than CMML. For AML: Acute Promyelocytic Leukemia (APL) or Isolated extramedullary disease.
* Eligible for an immediate allogenic stem cell transplant (alloSCT).
* Current active use of nicotine products including tobacco, nicotine patches or vaping products.
* Prior bone marrow transplant (BMT) within 6 months of date of consent; or transplanted patients who received the last dose of immunosuppressive therapies within 3 months of date of consent.
* Has active autoimmune condition requiring immunosuppressive treatment or is receiving immunosuppressive therapy for the treatment of autoimmune disorders, allergies, or other clinical symptoms. Systemic steroids <10 mg (milligrams) daily of prednisone equivalent are allowed; and intermittent use of bronchodilators or inhaled steroids, local steroid injections, topical steroids are allowed.
* Received treatment with chemotherapy, biologic therapy, or wide-field radiation within 14 days of consent. Exceptions for hydroxyurea: For CMML and AML participants, hydroxyurea may be continued up to 72 hours prior to first dose of STX-0712. Hydroxyurea will also be permitted for first cycle of STX-0712 treatment for participants with proliferative CMML or AML with high white blood count (WBC ≥25,000/µL).
* Received an investigational treatment within 30 days prior to dosing with STX-0712.
* Received Granulocyte Colony Stimulating Factor [G-CSF], Granulocyte Macrophage Colony Stimulating Factor [GM-CSF], erythropoietin, romiplostim, or other growth factors within 2 weeks prior to first dose of STX- 0712.
* Received a live or live attenuated vaccine within 30 days before the first dose of STX-0712.
* Clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association class 3 or 4 congestive heart failure, uncontrolled or unstable chest pain, history of heart attack(s), or stroke within 6 months prior to consent, uncontrolled high blood pressure, or clinically significant arrhythmias not controlled by medication).
* QT interval corrected by Fridericia's formula (QTcF) >470 msec for both men and women on Screening electrocardiogram(s) (ECG). Patients with a bundle branch block must have QT interval corrected for bundle branch block.
* Other than AML or CMML, active malignancy and/or cancer history that requires active therapy. Patients with the following neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ (including superficial bladder cancer), cervical intraepithelial neoplasia, or organ-confined prostate cancer with no evidence of progressive disease.
* Active, uncontrolled bacterial, fungal, or viral infection.
* Known human immunodeficiency virus (HIV).
* Active or chronic hepatitis B or hepatitis C infection.
* Evidence of any other severe or uncontrolled systemic diseases, any other serious and/or unstable pre-existing medical conditions, psychiatric disorder, or other conditions that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and/or minimum effective dose (MED) | Until the end of Dose Escalation (approximately 12 months)
  Incidence of dose-limiting toxicity (DLT) events during the DLT monitoring period

SECONDARY OUTCOMES:
To evaluate the overall safety and tolerability of STX-0712 | Until the end of the study (approximately 24 months)
  Incidence of adverse events (AEs), characterized overall and by type, seriousness, relationship to study treatment, timing, and severity graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
To evaluate the initial anti-tumor activity of STX-0712 in the CMML and AML cohorts | Until the end of the study (approximately 24 months)
  Investigator-assessed overall response rate (ORR) as measured by standard response criteria:
  For CMML: Proportion of participants achieving complete response (CR), complete cytogenetic remission, partial response (PR), marrow response, and clinical benefit according to the 2015 myelodysplastic/myeloproliferative neoplasms International Working Group (MDS/MPN IWG) criteria.
  For AML: Proportion of participants achieving complete remission (CR), CR with partial hematologic recovery (CRh), complete remission with incomplete count recovery (CRi), morphological leukemia-free state (MLFS), and PR according to modified European Leukemia Network (ELN) 2022 criteria
To evaluate the initial anti-tumor activity of STX-0712 in the CMML and AML cohorts | Until the end of the study (approximately 24 months)
  Absolute decrease in peripheral blood monocytes by 50% from baseline in CMML and AML.
Pharmacokinetics of STX-0712: maximum concentration (Cmax) | Until the end of the study (approximately 24 months)
  maximum concentration (Cmax)
Pharmacokinetics of STX-0712: time to reach maximum concentration (Tmax) | Until the end of the study (approximately 24 months)
  time to reach maximum concentration (Tmax)
Pharmacokinetics of STX-0712: area under the curve (AUC) | Until the end of the study (approximately 24 months)
  Area under the curve (AUC)
Pharmacokinetics of STX-0712: half-life (t½) | Until the end of the study (approximately 24 months)
  Half-life (t½)
To characterize the PD profile of STX-0712 after single and repeat-dose administration | Until the end of the study (approximately 24 months)
  Decrease in tumor cells following STX-0712 dose STX-0712 single-dose and repeat-dose blood PD biomarkers of target activation

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, MSc, MBA, Study Director — Solu Therapeutics
Locations (7):
- United States (7):
  - Stanford University, Stanford, California
  - Moffitt, Tampa, Florida
  - DFCI, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - OHSU, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
First-in-Human study using a first-in-class compound.